CLINICAL TRIAL: NCT05016115
Title: A Four-Year Longitudinal Study of Empathy Levels in Undergraduate Physiotherapy Students
Brief Title: Longitudinal Study of Empathy Levels in Physiotherapy Students
Acronym: Empathy
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Hulya Yucel, Assoc. Prof., Saglik Bilimleri Universitesi
Other Study IDs: 71306642/050-01-04/257
Record Dates: First submitted 2021-07-22; First posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Longitudinal Study of Empathy Levels in Physiotherapy Students
Keywords: empathy; longitudinal studies; students
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- physiotherapy students: Totally 120 physiotherapy students at a non-governmental university in Istanbul participated in this study.
  Interventions: Behavioral: survey

INTERVENTIONS:
Behavioral: survey — The Turkish reworded student version of the Jefferson scale of physician empathy was used. Empathy scores were compared related to study years and gender.

SUMMARY:
'Empathy' is a core term of occupations related to health sciences like physiotherapy. In physiotherapy education programs, empathy is necessary to have a successful cooperation with the clients. This study was planned to follow the changes of empathy levels in physiotherapy students of a four-year bachelor program and therefore enhance the curriculum related to the results. To the best of our knowledge, this research is the first longitudinal study about empathy levels of students in Turkey. Hypotheses: Empathy levels of the students increase year by year (1). Female students are more empathetic than male ones (2).

DETAILED DESCRIPTION:
Totally 120 physiotherapy students at a non-governmental university in Istanbul participated in this study. The Turkish reworded student version of the Jefferson scale of physician empathy was used. Empathy scores were compared related to study years and gender. Empathy scores relevant to gender were compared using Mann-Whitney U test. The Kruskal-Wallis one-way analysis of variance was used for differences among the four study years.

ELIGIBILITY:
Inclusion Criteria:

* attending the first through fourth year of physiotherapy department
* being willing to participate in the study

Exclusion Criteria:

do not continue in physiotherapy department

Ages: 19 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: physiotherapy students
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Empathy levels of the students | 5 minutes
  It was measured if the empathy levels of the students increase year by year

SECONDARY OUTCOMES:
Empathy levels of female students | 5 minutes
  It was measured if female students are more empathetic than male ones

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen PJ, Huang CD, Yeh SJ. Impact of a narrative medicine programme on healthcare providers' empathy scores over time. BMC Med Educ. 2017 Jul 5;17(1):108. doi: 10.1186/s12909-017-0952-x. PMID 28679379
- [Background] Hojat M, Gonnella JS. Eleven Years of Data on the Jefferson Scale of Empathy-Medical Student Version (JSE-S): Proxy Norm Data and Tentative Cutoff Scores. Med Princ Pract. 2015;24(4):344-50. doi: 10.1159/000381954. Epub 2015 Apr 28. PMID 25924560